CLINICAL TRIAL: NCT01487837
Title: A Phase IV, Randomized, Single Center, Parallel Group Trial of Human Fibrinogen Concentrate (Haemocomplettan) in the Treatment of Dilutional Coagulopathy During Major Pediatric Surgery
Brief Title: Fibrinogen for Treatment of Pediatric Dilutional Coagulopathy. FibPaed Study.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Children's Hospital, Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KEK-ZH-Nr. 2011-0440
Record Dates: First submitted 2011-12-05; First posted 2011-12-07 (Estimated); Last update posted 2014-10-27 (Estimated); Status verified 2014-10

CONDITIONS: Blood Coagulation Disorders; Hemorrhage
Keywords: Fibrinogen; Blood coagulation disorders; Postoperative bleeding; Transfusions
MeSH Terms: conditions — Blood Coagulation Disorders; Hemorrhage; Postoperative Hemorrhage

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fibrinogen if FibTEM < 8 mm (Active Comparator): Administration of fibrinogen concentrate if ROTEM FibTEM revealed MCF < 8 mm
  Interventions: Drug: Human fibrinogen concentrate
- Fibrinogen if FibTEM < 13 mm (Experimental): Administration of fibrinogen concentrate if ROTEM FibTEM revealed MCF < 13 mm
  Interventions: Drug: Human fibrinogen concentrate

INTERVENTIONS:
Drug: Human fibrinogen concentrate — Administration of human fibrinogen concentrate (30 mg / kg bw) over 15 min Repetition if hourly intraoperative ROTEM measurements revealed hypofibrinogenemia according to treatment group definition
  Other Names: Haemocomplettan P, CSL Behring

SUMMARY:
The purpose of this study is to compare two different thromboelastometry (ROTEM) trigger levels for administration of human fibrinogen concentrate (Haemocomplettan P) in the treatment of perioperative dilutional coagulopathy during major pediatric surgery. The study hypothesis is that administration of fibrinogen concentrate triggered by a ROTEM FibTEM MCF < 13 mm might reduce the total amount of transfused red cell concentrate during 24 hours after start of surgery as compared to a trigger level of ROTEM FibTEM MCF < 8 mm.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females
* Age 6 months to 17 years
* Scheduled for elective scoliosis surgery or major craniofacial surgery
* Written informed consent has been obtained
* Intraoperative hypofibrinogenemia according to definition of treatment groups

Exclusion Criteria:

* Preexisting congenital or acquired coagulation disorder
* Medical history of estimated increased bleeding tendency
* Ongoing coagulation therapy
* Clinical signs or diagnosis of acute thromboembolism
* Intolerance of study drug
* Participation at another clinical trial
* Pregnant or lactating women

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 57 (Actual)
Dates: Start 2012-01; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Total amount of transfused red cell concentrate | 24 hours after start of surgery

SECONDARY OUTCOMES:
coagulation measurements | 24 hours after start of surgery
  influence on viscoelastic coagulation measurements (ROTEM), plasmatic coagulation testing, FXIII levels, and endogenous thrombin potential
length of stay on PICU | 14 days after surgery or discharge of hospital, whatever occurs earlier
Additional transfusion/blood products requirements | 24 hours after start of surgery
Occurence of re-bleeding, surgical revision | 14 days after surgery or discharge of hospital, whatever occurs earlier
Occurence of (severe) adverse events | 14 days after surgery or discharge of hospital, whatever occurs earlier

CONTACTS AND LOCATIONS:
Overall Officials: Thorsten Haas, MD, Principal Investigator — Zurich University Children's Hospital
Locations (1):
- Zurich University Children's Hospital, Zurich, Switzerland

REFERENCES:
- [Derived] Restin T, Schmugge M, Cushing MM, Haas T. Comparison between intraoperative bleeding score and ROTEM(R) measurements to assess coagulopathy during major pediatric surgery. Transfus Apher Sci. 2021 Oct;60(5):103191. doi: 10.1016/j.transci.2021.103191. Epub 2021 Jun 19. PMID 34215519
- [Derived] Haas T, Spielmann N, Restin T, Seifert B, Henze G, Obwegeser J, Min K, Jeszenszky D, Weiss M, Schmugge M. Higher fibrinogen concentrations for reduction of transfusion requirements during major paediatric surgery: A prospective randomised controlled trial. Br J Anaesth. 2015 Aug;115(2):234-43. doi: 10.1093/bja/aev136. Epub 2015 May 15. PMID 25982134